CLINICAL TRIAL: NCT04103983
Title: An Investigation of the Efficacy of a Novel Sensory Discrimination Training Device for the Management of Phantom Limb Pain: A Randomised, Single-blind, Placebo-controlled Trial. [PHANTOM RELIEF Trial]
Brief Title: Sensory Retraining for Phantom Limb Pain
Acronym: PHANTOM RELIEF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Teesside University (Other)
Collaborators: 2PD Ltd (Unknown); Royal Commission for the Exhibition of 1851 (Unknown)
Responsible Party: Principal Investigator, Sarah Oatway, Clinical Trial Manager, Teesside University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2023 July 16692; 250337 (Other: IRAS)
Record Dates: First submitted 2019-09-20; First posted 2019-09-26 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Phantom Limb Pain
MeSH Terms: conditions — Phantom Limb

STUDY DESIGN:
Intervention Model Description: Randomised, single blind, controlled, mixed-methods study.
Who Masked: Participant, Outcomes Assessor
Masking Description: The participants and statistician will be blinded to treatment allocation. Outcome measures will be self reported by the participants. The care provider will not be blind, as they are required to provide specific instructions for each group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sensory Retraining Interactive Device (Active Comparator): The interactive device is a sensory retraining device. A pad consisting of twelve equally spaced electrodes is placed over the residual limb. This pad is connected to a handheld device which delivers an electrical current to the electrodes. The type of electrical current is similar to a TENS device. The device stimulates the skin via one of the electrodes, with either a single, or a rapid burst of pulse(s). The device touch screen then presents the questions, Which electrode (location) was stimulated? Was a single continuous or a rapid burst of pulses given (stimulation type)? The user responds via the screen and is told if they are correct. If correct, a new stimulus is delivered (different location and type) and the process repeated. If incorrect, the user is informed of the correct response, the same stimulation (location and type) is repeated once before moving onto to a new stimulus.
  Interventions: Device: Sensory retraining device
- Placebo Sensory Retraining Non-Interactive Device (Placebo Comparator): The placebo non-interactive device is physically visually identical to the interactive device. This device delivers the stimulation using microcurrents that the participants may or may not feel. There is no interaction required with this device i.e. there is no Q&A element, feedback nor response dependent progression.
  Interventions: Device: Sensory retraining device

INTERVENTIONS:
Device: Sensory retraining device — All participants will be given a device to keep at home and will be asked to use it for 60 minutes each day, as one block, or as multiple shorter sessions of 20 minutes minimum duration. Participants will be asked to use their device on 15 of the 21 days. They will be asked to spread out the use of the device over the 21 days. Participants are asked to record device use in a diary.

SUMMARY:
86-87% of people who have had an amputation still feel pain in the limb that has been amputated - Phantom limb pain (PLP). Sensory retraining is a form of treatment for PLP where a special form of electrical stimulation is delivered to the residual limb.

The theory is that this stimulation changes activity in the brain that helps to reduce the person's pain. Two new types of sensory retraining device for the treatment of phantom limb pain have been developed. One type requires the user to interact with the device while the other is a non-interactive device. Both devices are new so it is unknown as to how well they may work, or which is best, therefore both will be tested in this study.

This study will be undertaken remotely, using video call, telephone and email for communication. The study will compare the effect of both devices for efficacy. One hundred people with PLP will be recruited from the NHS and the general public and randomised to receive either the interactive or non-interactive device or their placebo equivalents. A health care professional will train the research participants how to use their device. Participants will then use their device at home for 3 weeks. To ensure that they are using their devices as required, the researchers will keep in contact throughout the three week treatment period, using a schedule of video calls, weekly phone calls and daily texts. Pain and function will be measured before treatment, after treatment and at a 3 month follow-up. Twelve participants will also be invited to a one-to-one interview to give their experience of the acceptability and usability of their device.

ELIGIBILITY:
Inclusion criteria

* Living in the UK
* All Genders
* Aged ≥18 years of age
* Women who self-declare:
* that they are post-menopausal, or permanently sterile*,

  - or -
* that it is physiologically impossible that they could be pregnant and not be aware they are.

Women who do not make one of the two declarations above, are only eligible if:

* they undertake a highly sensitive urine pregnancy test which is negative, prior (and as close in time as is possible) to beginning the treatment phase of the Trial,
* and -
* they agree to use a highly, or acceptably effective, contraceptive measure** during the treatment phase of the Trial.

  * fully healed residual limb (or stump) ***
  * single or multi limb amputation with the intervention applied to the participants limb of choice
  * experienced PLP rated as ≥4 on a 0-10 scale on at least 2 days in the week prior to enrolment
  * agree to inform us of the use of any new (to them) prescribed drug for their pain during the trial
  * any prescribed pharmacological treatment for the treatment of PLP stable for one month prior to commencing the trial , and agree not to undertake any non-pharmacological treatments for their PLP during the trial (e.g., mirror therapy)
  * agree to inform us of any other health care received related to the amputated limb during the trial (e.g., physiotherapy or occupational therapy) whether specific to PLP or not
  * any previous non-pharmacological PLP treatment must have terminated at least 1 month prior to commencing the trial
  * Participants will need access to a mobile smart phone and a device (laptop, iPad etc.) at home to receive text messages and take part in secure video conference calls and completion of online forms.

    *Post menopause is defined as no menses for 12 months without an alternative medical cause. Permanently sterile methods include hysterectomy, bilateral salpingectomy, and bilateral oophorectomy

    **Highly effective contraceptive methods being:
  * Combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation either oral, intravaginal, or transdermal
  * Progestogen only hormonal contraception associated with inhibition of ovulation, either oral, injectable, or implantable
  * Intrauterine device IUD
  * Intrauterine hormone-releasing system IUS
  * Sexual abstinence

Acceptably effective contraceptive methods being:

* Progestogen-only oral hormonal contraception, where inhibition of ovulation is not the primary mode of action
* Male or female condom with or without spermicide
* Cap, diaphragm or sponge with spermicide
* A combination of male condom with either cap, diaphragm or sponge with spermicide (double barrier methods)

  * Fully healed criteria: no bleeding, no oozing, no broken skin, no obvious sign of infection, such as swelling or redness, around the scar.

Exclusion criteria

* lacking Mental Capacity to give Informed Consent
* women who self-declare that they are pregnant, or that they will be trying to become pregnant, during the treatment phase of the Trial*
* impaired sensation as measured by hot/ cold test and sharp/ blunt test
* unable to read and speak English - the questionnaires being used have not been translated and validated in multiple languages and no facility is available to conduct nor translate/ back-translate semi-structured interview data
* epileptic
* active deep vein thrombosis, thrombophlebitis, or varicose veins
* fitted with a pacemaker
* has a metal implant in the area to be stimulated
* any residual limb complications such as cellulitis, wounds, infections etc.
* Active regions of known or suspected malignancy
* Any actively bleeding tissue or to persons with untreated haemorrhagic disorders
* Participating in any research trial of any intervention hypothesised to affect PLP
* Any current or recent history of substance misuse, alcohol, or drug dependency
* Any person, otherwise eligible, who commences any non-pharmacological treatment for PLP during the trial period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2024-02-09 (Actual); Primary Completion 2025-05-18 (Actual); Study Completion 2025-07-18 (Actual)

PRIMARY OUTCOMES:
The short form McGill Pain Questionnaire (SF-MPQ-2) | Day 1 (baseline prior to start) and Day 21 (end) of treatment period
  The primary outcome will be the total score of the McGill Pain Questionnaire revised (SF-MPQ-2)8 20 at the 3-week time point. The SF-MPQ-2 is a commonly used questionnaire to assess pain levels in a range of pain conditions. There are 22 items/ pain descriptors across 4 pain sub-scales/ domains: continuous, intermittent, neuropathic, and affective. Participants rate each item on an 11-point (0-10) scale, where 0 = none and 10 = worst possible pain. The mean of the 22 items provides the SF-MPQ-2 total score. Two or more missing responses on any sub-scale results in an invalid outcome. A targeted effect size of 1 unit difference between groups will be used.

SECONDARY OUTCOMES:
Overall Pain: Visual Analogue Scale (100mm): | Day 1 (baseline prior to start) and Day 21 (end) of treatment period and at 3 month follow up point post end of treatment
  Participants will be asked to rate their phantom limb pain over the last week using a pain visual analogue scale consisting of a 100mm line with anchor statements of 0 representing no pain and 100 the worst pain imaginable. The participant will be asked to place a mark through the line to represent their pain. Participants will be asked to record the number of phantom limb pain episodes they have experienced over the past week.
Frequency adjusted pain score: (0-100) | Day 1 (baseline prior to start) and Day 21 (end) of treatment period and at 3 month follow up point post end of treatment
  Participants will be asked to record the frequency of PLP episodes they have experienced over the past week from 1 = all the time to 5 = Once a day or less per week. The overall pain score will be divided by the frequency value to create a composite frequency adjusted pain score ranging from 0-100.
General Subjective Outcome Score (GSOS) | Day 21 (end) of treatment period and at 3 month follow up point post end of treatment
  Participants will be asked to rate their level of improvement Choosing one of six options, ranging from "a lot worse" to "completely better" (Harland et al. 2015).
The short form McGill Pain Questionnaire (SF-MPQ-2) | 3 month follow up point post end of treatment period
  The short form McGill Pain Questionnaire (SF-MPQ-2) (Dworkin et al, 2009):
  The short from McGill Pain Questionnaire (SF-MPQ-2) is a commonly used questionnaire to assess pain levels in a range of pain conditions. Twenty words which describe pain across the sensory, affective, evaluative and miscellaneous domains are presented to the participant who is asked to choose which word best describes their pain in the last week and to rate how intense that descriptor of pain was on a 0-10 scale.
Trinity Amputation and prosthetic evaluation scale (modified) (TAPES) | Day 1 (baseline prior to start) and Day 21 (end) of treatment period and at 3 month follow up point post end of treatment
  Participants will be asked to complete a modified version of the Trinity Amputation and prosthetics evaluation scale (TAPES scale).The TAPES has been modified in that it only asks about issues specific to PLP, residual limb (or stump) pain, and phantom sensations.
EQ5D5L | Day 1 (baseline prior to start) and Day 21 (end) of treatment period and at 3 month follow up point post end of treatment
  A brief easy to use validated measure of quality of life. The EQ5D contains five items related to mobility, self-care, usual activities, pain and anxiety/depression. It also contains a visual analogue scale for rating general health.
Sleep Disturbance | Day 1 (baseline prior to start) and Day 21 (end) of treatment period and at 3 month follow up point post end of treatment
  Participants will be asked to complete the PROMIS Short Form v.1.0 - Sleep Disturbance 4a questionnaire. This is a self-reported questionnaire reporting perceptions of sleep quality, sleep depth, and restoration associated with sleep. It assesses sleep disturbance over the past seven days. There are four questions, each containing a 5-point Likert Scale, ranging from Very Poor to Very Good. The questions are then combined to create a score out of 100 (Gershan et al. 2010).
Participant satisfaction | Day 21 (end) of treatment period and at 3 month follow up point post end of treatment
  Six item rating scale. Participants will be asked to answer the question,
  "How likely are you to recommend the device to other people who had phantom limb pain following an amputation?" by choosing one of six options, ranging from "extremely likely" to "extremely unlikely".
Device Usability | Day 21 (end) of treatment period
  After treatment, to investigate usability, all participants will be asked to rate how easy do you think the device was to use on a Visual Analogue Scale (VAS) (100mm) with 0 representing not at all easy to use and 100 representing extremely easy to use.
Study Diary (medication use/device use/pain levels) | Each Day Days 1 (baseline prior to start) to Day 21 (end) of treatment period and at 3 month follow up point post end of treatment
  Participants will be asked to report on their daily medication usage over the duration of the trial in a study diary. The participant will be sent a daily notification by the SMART-TRIAL platform to remind them to complete the study diary for the three week treatment period. The diary will ask for the frequency, dosage and class of medication taken each day. In addition, patients will be asked to rate their phantom limb pain on a scale from 0-10 each day, the frequency of those pain episodes, and to record how many minutes they used the device each day.
Concordance with Protocol | Each Day Days 1 (baseline prior to start) to Day 21 (end) of treatment period
  The frequency and duration of use of the SP1X device will be documented in the daily study diary and compared against the protocol that participants were asked to adhere to. This data will also be automatically captured by the device.
Credibility of Devices | At 3 month follow up point post end of treatment
  Participants will be asked Which of the following four devices do you think you received? 1. A real interactive device, 2. A sham/placebo interactive device, 3. A real non-interactive device or 4. A sham/placebo non-interactive device? And then How confident are you that your device was (form inserts answer 1,2,3 or 4) on a 0-100 scale with 0 being not at all confident and 100 being completely confident?

CONTACTS AND LOCATIONS:
Overall Officials: Cormac Ryan, Professor, Principal Investigator — Teesside University
Locations (1):
- Teesside University, Middlesbrough, Tees Valley, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Oatway S, Martin D, Graham A, Batterham A, MacSween A, Smith S, Ravindran D, Ryan C. Efficacy of a novel sensory discrimination training device for the management of phantom limb pain: protocol for a randomised placebo-controlled trial. BMJ Open. 2025 Nov 9;15(11):e101657. doi: 10.1136/bmjopen-2025-101657. PMID 41213687

DOCUMENTS (1):
  • Statistical Analysis Plan (2024-09-04): https://cdn.clinicaltrials.gov/large-docs/83/NCT04103983/SAP_000.pdf